CLINICAL TRIAL: NCT04868448
Title: Cohort Study to Measure COVID-19 Vaccine Effectiveness Among Health Workers in Georgia
Brief Title: COVID-19 Vaccine Effectiveness Among Health Workers in Georgia
Acronym: COV19HWVE_GE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Disease control and Public Health (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Dr.Lia Sanodze, Principal Investigator, National Center for Disease control and Public Health
Other Study IDs: CERC.0097B
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: Vaccine effectiveness; Health workers; Georgia; Cohort study
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccinated participants: Participants who received 1or 2 doses of the Covid-19 vaccines
  Interventions: Biological: Covid-19 vaccines
- Unvaccinated participants: Participants who have not received any dose of the Covid-19 vaccines

INTERVENTIONS:
Biological: Covid-19 vaccines — Observation of individuals who received one or more doses of covid-19 vaccines.
  Groups: Vaccinated participants

SUMMARY:
This is a prospective one-year cohort study of hospital-based health workers in Georgia to evaluate the effectiveness of COVID-19 vaccine in preventing laboratory-confirmed SARS-CoV-2 infection and COVID-19 disease.

DETAILED DESCRIPTION:
Many critical questions remain about the effectiveness of COVID-19 vaccines in real-world settings. These questions can only be answered in post-introduction vaccine effectiveness studies.

This is a prospective one-year cohort study of hospital-based health workers in Georgia to evaluate the effectiveness of COVID-19 vaccine in preventing laboratory-confirmed SARS-CoV-2 infection and COVID-19 disease. Health Workers (HWs) are the target population in this study because they have been prioritized to be the first group to receive the vaccine in Georgia and offer an early opportunity to evaluate the vaccine in a population in which it is critical that an effective vaccine be deployed.

HWs should be enrolled after the study protocol is approved by the local ethical review committee. All HWs eligible to be vaccinated with COVID-19 vaccine can be enrolled in the study, including those who intend to get vaccinated, those who do not plan on getting vaccinated, and those who are not sure. For HWs who have already been vaccinated at enrolment, priority will be given to those who have received their first COVID vaccine no more than 4 days prior to the date of enrolment. The target enrolment is 1600 participants.

At enrolment, study participants will complete a baseline enrolment survey about demographics, clinical comorbidities, and work and community-related behaviors related to infection risk, and recent symptoms. In addition, a baseline serology will be collected from participants at enrolment.

For study participants who have not received their first COVID-19 vaccine at enrolment but receive their first vaccine 14 days or more after enrolment, an additional blood sample will be collected. In addition, a brief symptom questionnaire about recent symptoms will be administered.

During the course of the study, participants will be actively followed for suspected COVID-19 infection. Participants will be asked to complete weekly symptom questionnaires to screen for clinically significant COVID-19. Participants who meet a suspected case definition, defined according to the Georgian national case definition should provide a respiratory sample which will be collected by trained HW. Respiratory specimens will be tested for SARS-CoV-2 by RT-PCR.

All or subset of positive samples from study participants will undergo genetic sequencing, resources permitting.

Finally, after 3, 6, 9 and 12 months of the study, as resources permit, serology will be collected from participants. Serology will be tested for antibodies to SARS-CoV-2 by tests for vaccine-induced antibodies and antibodies that result from natural infection.

Vaccine effectiveness should be analysed as described in the analysis section below.

In addition to the final analysis at the end of the one-year period, interim quarterly (every three months) analyses will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

All HWs eligible to receive the COVID-19 vaccination according to the national guidelines of Ministry of Health (MoH).

* HWs working at Batumi Republican Clinical Hospital, Vakhtang Bochorishvili Clinic, Academician N. Kipshidze Central University Clinic, Bokeria Tbilisi Referral Hospital, Caucasus Medical Centre, and Infectious Diseases and AIDS Center.
* HWs who have already been vaccinated with a single dose of vaccine against COVID-19 as part of the early COVID-19 vaccine rollout can be included.

Exclusion Criteria:

* HWs who are not eligible for COVID-19 vaccination or have a contraindication to vaccination should not participate in the study.
* HWs who do not work at above mentioned hospitals
* HWs under 18 years of age.
* HWs who have already been vaccinated with two doses of vaccine against COVID-19 before enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of health workers in the above hospitals, eligible for vaccination, with no contraindication to receive COVID-19 vaccine. HWs include all categories of staff working in the hospitals, including clinical and non-clinical/administrative staff and staff with direct patient interaction and those without direct patient interaction. All HWs at the above hospitals who are eligible for vaccination, according to Ministry of Health guidelines, will be eligible for enrolment, regardless of their intention to receive the COVID-19 vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Covid-19 vaccine effectiveness | 12 months
  any SARS-CoV-2 laboratory confirmation by RT-PCR in an asymptomatic, or symptomatic patient

CONTACTS AND LOCATIONS:
Overall Officials: Khatuna C Zakhashvili, MD, Principal Investigator — National Center for Disease control and Public Health
Locations (6):
- Georgia (6):
  - The Batumi Republican Clinical Hospital, Batumi, Adjara
  - The Bokeria Tbilisi Referral Hospital, Tbilisi
  - Academician N. Kipshidze Central University Clinic, Tbilisi
  - The Bochorishvili Clinic, Tbilisi
  - The Infectious Diseases and AIDS Center, Tbilisi
  - The Caucasus Medical Centre, Tbilisi

IPD SHARING:
Plan to Share IPD: No